CLINICAL TRIAL: NCT05579470
Title: Expanding Medication-Assisted Therapies in Central Asia
Acronym: ExMAT CA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Den Sooluk Nuru (Unknown); Institute for International Health and Education (Unknown); Global Health Research Center of Central Asia (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000031029; 1R01DA054851-01A1 (NIH)
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder
Keywords: HIV; OUD; OAT; Central Asia
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: THe investigators propose a quasi-experimental, pretest-posttest design to evaluate the effect of the NIATx strategy on OAT scale-up for three CA countries. Specifically interested in assessing how the introduction of a NIATx model affects two primary outcomes: (1) rate of entry onto OAT, and (2) retention on OAT. Though the implementation science field is rapidly evolving, such an approach is limited by its assumption that existing data were collected and recorded in a manner that adheres to the fidelity of the measures - a noted innovation in this proposal. This limitation is addressed prospectively recording OAT entry and attrition over an extended time period (36 months) and, as part of Aim 3, collect inner and outer context and bridging and innovation of EBP factors as repeated measures to examine trajectories and factors that are associated with them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NIATx Model (Other): Receiving NIATx Coaching
  Interventions: Behavioral: NIATx

INTERVENTIONS:
Behavioral: NIATx — For each country, the learning collaborative will be comprised of a Chief Narcologist from each region where the investigators will initially train them and the coaches using all the tools from the NIATx Academy (2-3-day training). The national coach for each country will receive ongoing and in-depth coaching from a US-based super coach. A nationwide Nominal Group Technique (NGT) will be conducted to assess barriers and potential targets to guide decision-making about changes. At the end of the initial meeting, each Chief Narcologist (CN) will be able to identify a change target for Plan, Do, Study, Act (PDSA) (entry, retention) and create a Change Project Form to state what will be done (e.g. flowcharting), who is involved (team), what are the measures and timeframe (<4 weeks).

SUMMARY:
Central Asia (CA) represents the most rapidly growing HIV epidemic region worldwide, concentrated in people who inject drugs (PWID) and their sexual partners, and scaling up opioid agonist therapies (OAT) in this region is the most cost-effective strategy to prevent new HIV infections, and more effective when combined with antiretroviral therapy (ART). The investigators propose to use the Network for the Improvement of Addiction Treatment (NIATx) implementation strategy to scale-up OAT in three diverse Central Asian countries (Kazakhstan, Kyrgyzstan, Tajikistan) and guided by the Exploration-Planning-Implementation-Sustainment (EPIS) framework. Understanding the trajectories of implementation and scale-up in this context may emerge through creating communities of practice, especially when cohesion and competence evolves, and may guide other healthcare delivery challenges in the region (e.g., HIV, TB); as well as build important regional expertise and understanding implementation trajectories should help support OAT program sustainability.

DETAILED DESCRIPTION:
Central Asia (CA) represents the most rapidly growing HIV epidemic region worldwide, concentrated in people who inject drugs (PWID) and their sexual partners. Scaling up opioid agonist therapies (OAT) in CA is the most cost-effective strategy to prevent new HIV infections, and more effective when combined with antiretroviral therapy (ART). OAT, when adequately scaled, controls HIV epidemics through both primary and secondary prevention (increased engagement along the entire HIV treatment cascade). CA countries have especially low OAT (and ART) coverage and are uniquely impacted by their proximity to opioid trade routes, a myriad of patient, provider, healthcare and policy barriers and suboptimal implementation. CA countries share a similar Semashko healthcare system, but differ by political, cultural and economic trajectories since independence from the Soviet Union. Such healthcare systems are especially challenging for implementation of evidence-based practices (EBPs). Moreover, the HIV treatment cascade differs in Kazakhstan (KZ), Kyrgyzstan (KY) and Tajikistan (TJ) with low levels of HIV testing (71%, 61% and 48%), being on ART (~30%) and viral suppression (20%, 18%, 22%), respectively. OAT coverage is similarly low (0.2%, 4.6% and 2.8%) for the 120,500, 25,000 and 22,500 PWID, respectively. The investigators propose to use the Network for the Improvement of Addiction Treatment (NIATx) implementation strategy to scale-up OAT in three diverse CA countries guided by the Exploration-Planning-Implementation-Sustainment (EPIS) framework.

Using the investigators experiences with NIATx to scale-up OAT in Ukraine, the EPIS framework will be used where the investigators will first assess the barriers and facilitators to OAT scale-up, including inner and outer context and bridging factors associated with OAT innovations as part of exploration/preparation. Despite its unequivocal efficacy, it was perceived as negative by both patients and providers in Ukraine. Myths surrounding OAT combined with structural factors within clinics accounted for 82% of the barriers. The investigators then implemented NIATx by training in-country coaches and used a menu of tools and quality improvement techniques to scale-up OAT to increase OAT entry and retention. EPIS relies on dynamic use of implementation to adapt to the context. Collaborative learning is key feature of NIATx that involves a transformation to adoption and scale-up of EBPs. OAT implementation, however, requires adaptation of implementation strategies to local contextual factors, including available resources, expertise, and cultural norms, which must be accomplished for successful implementation. Such adaptation, however, must be understood to promote sustainability and to install promising practices that are unique to the context. Health delivery in CA is based on vestiges of Soviet-era Semashko health systems which are siloed, rigidly vertical and do not promote teamwork. Observations from Ukraine suggest that group cohesion may emerge through collaborative learning, but it is not linear and outcomes among group members differ. Understanding the trajectories of implementation, a core feature of EPIS, may in this context emerge through creating communities of practice, especially when cohesion evolves, and may guide other healthcare delivery challenges in the region (e.g., HIV, TB). Using NIATx to build important regional expertise and understanding implementation trajectories should help support OAT program sustainability. The specific aims are:

1. To create a socio-ecological framework for OAT delivery by conducting formative research to assess client-level, program-level and structural facilitators and barriers to entry into and retention in OAT in each country in order to create improved, sustainable models of OAT delivery that are contextually relevant, including integration of OAT into primary and HIV clinical care settings.
2. To scale-up OAT in 3 diverse Central Asian countries by training and coaching national experts in Kazakhstan (KZ), Kyrgyzstan (KG) and Tajikistan (TJ) on the use of NIATx.
3. To use latent class growth analyses to identify implementation trajectories of OAT, scale-up using NIATx in the Eastern Europe and Central Asia (EECA) context and explore which organizational, professional and group dynamic characteristics are associated with these trajectories and related to individual level outcomes (i.e., OAT scale-up).

As part of the implementation and sustainability plan, and consistent with NIATx, the investigators will convene stakeholder meetings to bridge inner (National and Oblast Chief Narcologists) and outer (e.g. Non-Governmental Organization (NGOs), Ministry of Health, external funders and experts) factors to guide initial implementation, review findings from the investigators studies and use information to inform policies for expanding OAT in each CA country. These meeting will inform implementation and guide structural policy changes to promote sustainability. Significance is high given CA having the most rapidly evolving HIV epidemic worldwide, concentrated in PWID and their sexual partners and where current implementation efforts have failed. Innovation is high by using NIATx and its extensive toolkit to facilitate OAT scale-up alongside an in-depth assessment of key NIATx elements that contribute to success in this context. Success is likely to be high given the experience of the US and Central Asian teams, their previous collaborative research and a common goal to control HIV in the region. Public health benefit is likely to be high given the need to simultaneously address both treatment and prevention of HIV and opioid use disorder (OUD).

ELIGIBILITY:
Inclusion Criteria:

i. Aim 1: The inclusion criteria for Aim 1 Consists of:

1. Quantitative surveys for PWID

   1. 18 years or older
   2. Meeting DSM-V criteria for opioid dependence
   3. Be either treatment naïve and seeking OAT or be on OAT for < 90 days
2. Organizational Assessments for OAT Delivery Staff

   1. 18 years or older
   2. Currently working as an OAT delivery professional at an OAT delivery site
3. Focus Groups (PWID on OAT)

   1. 18 years or older
   2. Meeting DSM-V criteria for opioid dependence
   3. Be either treatment naïve and seeking OAT or be on OAT for < 90 days
4. Focus Groups (PWID not on OAT)

   1. 18 years or older
   2. Meeting Diagnostic and Statistical Manual of Mental Disorders(DSM)-V criteria for opioid dependence
   3. Be OAT naïve (defined as never having been on OAT or having not received treatment for > 1 year)
5. Focus Groups (OAT delivery staff)

   1. 18 years or older
   2. Currently working as an OAT delivery professional at an OAT delivery site

ii. Aim 2: The inclusion criteria for Aim 2 consists of:

1. 18 years or older
2. Currently assigned as a Chief Narcologist for an Oblast

iii. Aim 3: The inclusion criteria for Aim 3 consists of:

1. 18 years or older
2. Authorized as a professional to work at an OAT delivery site

Exclusion Criteria:

* Not willing to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
OAT Census | 36 months
  Absolute number of patients on OAT per country
OAT Census per Oblast | 36 months
  Absolute number of patients on OAT per oblast

SECONDARY OUTCOMES:
New Patients | 36 months
  Total number of newly enrolled patients into OAT services, per country
New Patients per Oblast | 36 months
  Total number of newly enrolled patients into OAT services, per oblast
Dropout | 36 months
  Total number of patients dropping out of OAT services, per country
Dropout per Oblast | 36 months
  Total number of patients dropping out of OAT services, per oblast

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L Altice, MD, Principal Investigator — Yale University
Locations (4):
- Yale University, New Haven, Connecticut, United States
- Columbia University Global Health Research Center of Central Asia, Almaty, Kazakhstan
- Den Sooluk Nuru, Bishkek, Kyrgyzstan
- Institute for International Health and Education, Dushanbe, Tajikistan

IPD SHARING:
Plan to Share IPD: No